CLINICAL TRIAL: NCT02548780
Title: Pharmacokinetic Study in Patients With Unresectable Hepatocellular Carcinoma (HCC) Receiving Treatment With LifePearl Microspheres Loaded With Doxorubicin
Brief Title: LifePearl-Doxo Pharmacokinetic (PK) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T125E2
Record Dates: First submitted 2015-08-27; First posted 2015-09-14 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: HCC; Hepatocellular Carcinoma
Keywords: unresectable
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoembolization + Pharmacokinetics (Experimental): First cohort: Chemoembolization with Doxorubicin-loaded LifePearl™ microspheres (TACE): Escalation of dose loaded in microspheres from 75 mg to 150 mg. Pharmacokinetic testing in all patients.
  Second cohort: Chemoembolization with doxorubicin-loaded LifePearl™microspheres: microspheres loaded with maximum tolerated dose as established with dose escalation arm. Pharmacokinetic testing in all patients.
  Interventions: Device: Chemoembolization; Other: Pharmacokinetics

INTERVENTIONS:
Device: Chemoembolization — First, an angiography of the celiac trunk, superior mesenteric artery and hepatic artery will be obtained by using a peripheral arterial approach.
  Arterial embolization will be performed through catheterization of intrahepatic arteries, as selectively as possible (tumor feeders, subsegmental, segmental). The size of the microcatheter must be consistent with the size of LifePearl beads used. Microspheres of 200 µm will be be used. They will be loaded with the appropriate dose of doxorubicin injectable solution, mixed with the contrast media and distributed according to the location of the HCC lesions. The endpoint of the procedure will be achieved end when stasis of the feeders is achieved and confirmed with angiography of the whole liver.
  Other Names: Chemoembolization with LifePearl™ loaded with Doxorubicine
Other: Pharmacokinetics — Pharmacokinetic analysis will be performed in cohort I and II after the first treatment only. In addition to blood samples taken for biochemistry and haematology analysis, blood will be taken for pharmacokinetic assessment: Whole venous blood samples (6 ml in 2 tubes) will be taken from peripheral blood into ethylenediaminetetraacetic acid (EDTA) tubes prior to and at 5mins, 20mins, 40mins, 1h, 2h, 6h, 24h, 48h and 7 days after the procedure, and if needed (i.e. value at d7 is detectable) at 1 month (for safety assessment visit) either during hospital stay or in the outpatient clinic.

SUMMARY:
The primary purpose of the study is to evaluate the pharmacokinetic profile, safety, and efficacy of LifePearl™ microspheres loaded with Doxorubicin in the treatment of unresectable HCC.

DETAILED DESCRIPTION:
This is a multicentre, prospective dose escalation/PK study, designed to assess the clinical performance of LifePearl™ beads loaded with Doxorubicin in the primary treatment of unresectable HCC by chemoembolization. Data from this study will be used as supportive data post CE-mark approval.

The main objective of the study is to evaluate the safety and pharmacokinetic profile of LifePearl™ beads loaded with Doxorubicin in the treatment of patients with unresectable liver cancer (HCC) by chemoembolization. This will be measured as treatment-related complications and plasma levels of Doxorubicin in peripheral blood.

In addition, objective tumour response will be assessed by computed tomography or MRI.

Two cohorts of patients will be evaluated:

Cohort I to assess safety (dose escalation) and pharmacokinetic profile; Cohort II will assess pharmacokinetic profile, safety and efficacy with the doxorubicin dose determined with Cohort I.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* HCC diagnosed according to updated American Association for the Study of Liver Diseases (AASLD) or EASL-European Organization for Research and Treatment of Cancer (EORTC) criteria
* BCLC B patients or BCLC A patients not candidates for curative treatment (resection, transplantation, ablation) or who have failed/recurred after resection/ablation
* Tumor burden (located in one or two lobes) that can be sufficiently and selectively embolized with required dose of LifePearl loaded with doxorubicin
* Performance status (PS) 0
* Normal liver or compensated cirrhosis with preserved liver function (Child-Pugh A, score ≤ 6 points) without ascites in the absence of diuretic treatment
* Total bilirubin ≤2.0 mg/dl
* Adequate renal function (serum creatinine < 1.5 X ULN)
* Patient has provided written informed consent
* Patient is affiliated to social security or equivalent system (France only)

Exclusion Criteria:

* Patient previously treated with any intra-arterial therapy for HCC or sorafenib
* Eligible for curative treatment (resection/radiofrequency ablation (RFA), transplantation therapies);
* Advanced liver disease: Child-Pugh's B-C class or active gastrointestinal bleeding, encephalopathy. Bilirubin levels >2.0 mg/dl;
* Advanced tumoral disease: BCLC class C (vascular invasion -even segmental, extra-hepatic spread or cancer-related symptoms=PS of 1-2) or D class (WHO performance status 3 or 4)
* Patient with another primary tumor
* Patient with refractory ascites or on diuretic treatment
* Patient with history of biliary tree disease or biliary dilatation
* Portal vein thrombosis, porto-systemic shunt, hepatofugal blood flow or absent portal blood flow in the liver area to be treated
* Contraindication to multiphasic CT and MRI (e.g. allergy to contrast media);
* Any other contraindication for embolization or local doxorubicine treatment;
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Pregnant or breast-feeding women
* Patient is under judicial protection (France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Doxorubicine | 1 month
  Adverse Events (CTCAE v4.03 toxicity criteria) occurring within 28 days of the treatment. Grade ≥4 or Grade 3 in two patients at any one dose will mean the MTD has been achieved.
Peak Plasma Concentration (Cmax) | 1 month
  Maximum Plasma Concentration Doxorubicine
Adverse Events | 1 month
  Occurence of grade 3-4-5 treatment-related adverse events as Assessed by CTCAE v4.0.
Area under the Curve (AUC) | 1 month

SECONDARY OUTCOMES:
Angiographic Stasis | 1 day
  Ability to achieve stasis of bloodflow in the embolised arteries by angiographic assessment.
Total dose delivered | 2 months
  Sum of all doses Doxorubicine administered (maximum two chemoembolizations)
Response rate | 3 months
  Response rate assessed by Response Evaluation Criteria in Solid Tumors(RECIST) 1.1, EASL (European Association for the Study of the Liver) and mRECIST (modified RECIST) criteria 3 months after the first treatment
Time to Progression | 24 months
  Progression will be defined by the Barcelona Clinic Liver Cancer (BCLC)-refined RECIST
Overall Survival | 24 months
  The length of time from either the date of diagnosis or the start of treatment that patients diagnosed with the disease are still alive.
Progression Free Survival | 24 months
  The length of time during and after the treatment that a patient lives with the disease but it does not get worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Bruix, MD, Principal Investigator — CLÍNIC BARCELONA Hospital Universitari, Spain
Locations (3):
- Evgenidio Therapeftirio "Agia Trias", Athens, Greece
- Hospital Clínic i provincial de Barcelona, Barcelona, Spain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland